CLINICAL TRIAL: NCT00977392
Title: The Potential Role of Self-sampling in Women Who do Not Attend for Cervical Screening - a Randomised Controlled Trial
Brief Title: Self-Sampling in Women Who Do Not Undergo Routine Cervical Screening
Status: Completed | Type: Observational
Sponsor: Barts and the London School of Medicine and Dentistry (Other)
Organization: National Cancer Institute (NCI) (NIH)
Other Study IDs: CRUK-Westminster-Self-Sampling; CDR0000648274 (Registry Identifier: PDQ (Physician Data Query)); ISRCTN40182307 (Registry Identifier: ISRCTN (International Standard Randomised Controlled Trial Number Register)); EU-20963
Record Dates: First submitted 2009-09-12; First posted 2009-09-15 (Estimated); Last update posted 2013-08-07 (Estimated); Status verified 2009-09

CONDITIONS: Health Status Unknown; Precancerous Condition
Keywords: human papilloma virus infection; health status unknown
MeSH Terms: conditions — Precancerous Conditions; Papillomavirus Infections | interventions — Vaginal Smears; Early Intervention, Educational; Colposcopy

INTERVENTIONS:
Behavioral: compliance monitoring
Other: cervical Papanicolaou test
Other: educational intervention
Other: screening questionnaire administration
Other: survey administration
Procedure: colposcopy

SUMMARY:
RATIONALE: Women who do not undergo routine cervical screening may be more likely to collect a self-sample for human papillomavirus testing.

PURPOSE: This randomized clinical trial is studying self-sampling in women who do not undergo routine cervical screening.

DETAILED DESCRIPTION:
OBJECTIVES:

* To ascertain whether women who do not attend for cervical screening are more likely to respond to the opportunity to collect a self-sample for human papillomavirus (HPV) testing, or to respond to a further invitation to undergo a cervical smear.
* To ascertain whether such women will attend for further investigation if they have a positive screening test (HPV test or cervical smear).

OUTLINE: Patients are randomized to 1 of 2 arms.

* Control: Patients receive an invitation for a routine cervical smear and a cervical screening survey. Information regarding attendance for smear or colposcopy is collected at the Primary Care Trust.
* Study (self-sampling kit): Patients receive an explanatory letter, an information sheet about the study, a consent form, information about human papillomavirus (HPV) and HPV testing, a self-sampling test kit, and an invitation to take their own HPV sample and return it to the research group for processing. Patients also receive a cervical screening survey. Patients who attend for further investigation following a positive HPV result go to St. Mary's Hospital Colposcopy Unit, Paddington. During this visit cervical smear tests are performed and women are offered immediate colposcopy so that they would not need to return for colposcopic examination if their smear test is abnormal.

This study is peer reviewed and funded or endorsed by cancer research UK.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Women in Westminster Primary Care Trust (PCT) area eligible for routine cervical screening who have not responded to two invitations to attend for smears
* No women who have written to the PCT to document their refusal to take part in the National Health Service Cervical Screening Program (NHSCSP)
* No women who are not due for routine screening as part of the NHSCSP

PATIENT CHARACTERISTICS:

* Not pregnant
* Have been sexually active

PRIOR CONCURRENT THERAPY:

* No prior total abdominal hysterectomy

Min Age: 25 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 3000 (Estimated)
Dates: Start 2009-06; Primary Completion 2010-02 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Comparison of the percentages of women responding to the invitation to return a self-sampling kit vs responding to an invitation for a cervical smear

SECONDARY OUTCOMES:
Response to the invitation for further investigation following a positive test result (colposcopy for women with a smear showing mild dyskaryosis or above, smear +/- colposcopy for those with a positive HPV test)
Response to the request to return a survey regarding demographic information and reasons for previous non-attendance for screening

CONTACTS AND LOCATIONS:
Overall Officials: Anne Szarewski, MD, Principal Investigator — Queen Mary University of London
Locations (1):
- Barts and the London School of Medicine, London, England, United Kingdom

REFERENCES:
- See also: HPV self-sampling as an alternative strategy in non-attenders for cervical screening - a randomised controlled trial. Br J Cancer. 2011 Mar 15;104(6):915-20. doi: 10.1038/bjc.2011.48. Epub 2011 Feb 22. — http://www.ncbi.nlm.nih.gov/pubmed/21343937